CLINICAL TRIAL: NCT04443010
Title: A Study to Evaluate the Safety and Efficacy of the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF Plus Standard Temozolomide Chemoradiotherapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: Safety and Efficacy of L19TNF Plus Temozolomide Chemoradiotherapy in Patients With Newly Diagnosed Glioblastoma
Acronym: GLIOSUN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFTMZ-01/20
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: Open label phase I/II study in subjects with newly diagnosed glioblastoma. The study will be conducted in three consecutive parts: (i) first the dose finding part to determine the RD of L19TNF in combination with chemoradiotherapy, (ii) followed by a signal seeking part that investigates first signs of activity and (iii) then an activity evaluation part that studies the efficacy of L19TNF in combination with chemoradiotherapy against chemoradiotherapy alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 part: Dose Finding (Experimental): Patients will be treated in cohorts according to a 3+3 study design with standard treatment (consisting of radiotherapy of 60 Gy/30 fractions for 6 weeks plus 75 mg/m2 TMZ (temozolomide) daily (chemoradiotherapy), followed by 4 weeks of treatment break, followed by maintenance treatment with 6 maintenance cycles of TMZ 150-200 mg/m2 on Days 1 to 5 q28) combined with L19TNF at different dose levels on Day 1, 3, 5, 22, 24 and 26 of chemoradiotherapy and on Day 1, 3 and 5 of each 28-day chemotherapy maintenance cycle.
  Interventions: Drug: Onfekafusp alfa
- Phase 2 part: Signal Seeking (Experimental): 32 patients will receive standard chemoradiotherapy and L19TNF at RD and with the administration scheme established in phase I part of the study.
  Interventions: Drug: Onfekafusp alfa
- Phase 2b part: Activity Evaluation_control arm (Active Comparator): Patients will be randomized 1:1 and treated with either standard chemoradiotherapy and L19TNF as established in phase I part and the phase II part of this study or only chemoradiotherapy (control).
  - Arm 2: Patients will receive radiotherapy and TMZ (temozolomide).
  Interventions: Drug: Temozolomide
- Phase IIb part: Activity Evaluation_treatment arm (Experimental): Patients will be randomized 1:1 and treated with either standard chemoradiotherapy and L19TNF as established in phase I part and the phase II part of this study or only chemoradiotherapy (control).
  - Arm 1: Patients will receive radiotherapy, TMZ (temozolomide) and L19TNF.
  Interventions: Drug: Onfekafusp alfa; Drug: Temozolomide

INTERVENTIONS:
Drug: Onfekafusp alfa — This is an open label phase 1/2/2b study in subjects with newly diagnosed glioblastoma.
  The study will be conducted in three consecutive parts: First the dose finding part to determine the RD of L19TNF in combination with chemoradiotherapy, followed by a signal seeking part that investigates first signs of activity and then an activity evaluation part that studies the efficacy of L19TNF in combination with chemoradiotherapy against chemoradiotherapy alone.
  Other Names: L19TNF
  Arms: Phase 1 part: Dose Finding; Phase 2 part: Signal Seeking; Phase IIb part: Activity Evaluation_treatment arm
Drug: Temozolomide — Patients will receive radiotherapy and TMZ. Treatment start with chemoradiotherapy is foreseen after surgical resection or biopsy of glioblastoma
  Other Names: TMZ
  Arms: Phase 2b part: Activity Evaluation_control arm; Phase IIb part: Activity Evaluation_treatment arm

SUMMARY:
The purpose of this study is to explore the safety profile and establish a recommended dose (RD) for phase II of the antibody-cytokine fusion protein L19TNF plus standard TMZ chemoradiotherapy in patients with newly diagnosed glioblastoma.

The study will be conducted in three consecutive parts: a dose finding part to determine the RD of L19TNF in combination with chemoradiotherapy, followed by a signal seeking part that investigates first signs of activity and then an activity evaluation part that studies the efficacy of L19TNF in combination with chemoradiotherapy against chemoradiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18.
2. Patients with histologically confirmed newly diagnosed glioblastoma.
3. Karnofsky Performance Score (KPS) ≥ 70%
4. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
5. Female patients: negative pregnancy test for women of childbearing potential (WOCBP)* within 14 days of starting treatment. WOCBP must agree to use, from the screening to 6 months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.
6. Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required.
7. Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
8. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

   * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).

Exclusion Criteria:

1. Prior treatment for glioma, except surgery.
2. Inability to undergo contrast-enhanced MRI.
3. Intent to be treated with tumor-treating fields prior to progression.
4. Known history of allergy to TNF or TMZ, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
5. Absolute neutrophil count (ANC) < 1.5 x 10^9/L, platelets < 100 x 10^9/L or haemoglobin (Hb) < 9.0 g/dl.
6. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
7. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 2.0 x ULN).
8. INR > 1.5 ULN.
9. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
10. Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent.
11. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
12. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
13. Clinically significant cardiac arrhythmias or requiring permanent medication.
14. Abnormal LVEF or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator. Subjects with current or a history of QT/QTc prolongation are excluded.
15. Uncontrolled hypertension.
16. Known arterial aneurism at high risk of rupture.
17. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
18. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders.
19. Anxiety ≥ CTCAE Grade 3.
20. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
21. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 3 weeks of administration of study treatment.
22. Known history of tuberculosis.
23. Pregnancy or breast feeding.
24. Requirement of chronic administration of high dose corticosteroids or other immunosuppressant drugs. Subjects must have been either off corticosteroids, or on a stable or decreasing dose ≤ 4 mg daily dexamethasone (or equivalent) for 7 days prior to start of chemoradiotherapy. Limited or occasional use of corticosteroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
25. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
26. Concurrent malignancies unless the patient has been disease-free without intervention for at least 2 years.
27. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
28. Serious, non-healing wound, ulcer, or bone fracture.
29. Requirement of concurrent therapy with anticoagulants at therapeutic doses.
30. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
31. Any recent live vaccination within 4 weeks prior to treatment or plan to receive vaccination during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
For Phase 1: DLT | For Cohort 1 and Cohort 2 from Day 1 to Day 28 of the maintenance cycle; for Cohort 3, 4 and 5 from Day 1 to Day 42 of the chemoradiotherapy.
  Occurrence of dose limiting toxicity (DLT) assessed by frequency and grade of adverse events (AE) according to CTCAE v.5.0.
For Phase 2: Overall Survival | From beginning of treatment to 52 weeks
  Overall survival (OS) rate

SECONDARY OUTCOMES:
PFS | From the date of enrollment to the date of progression or death for any cause, whichever came first, assessed up to 58 weeks
  Progression Free Survival (PFS) will be assessed for all enrolled subjects.
ORR in CR | At week 10, at week 22, at week 34, at week 46 and at week 58
  Objective Response Rate (ORR): ORR is defined as the rate of patients with complete response (CR) (defined according to iRANO criteria)
ORR in PR | At week 10, at week 22, at week 34, at week 46 and at week 58
  Objective Response Rate (ORR): ORR is defined as the rate of patients with partial response (PR) (defined according to iRANO criteria)
DCR in CR | At week 10, at week 22, at week 34, at week 46 and at week 58
  Disease Control Rate (DCR) is defined as the rate of patients with complete response (CR) (defined according to iRANO criteria)
DCR in PR | At week 10, at week 22, at week 34, at week 46 and at week 58
  Disease Control Rate (DCR) is defined as the rate of patients with partial response (PR) (defined according to iRANO criteria)
DCR in SD | At week 10, at week 22, at week 34, at week 46 and at week 58
  Disease Control Rate (DCR) is defined as the rate of patients with stable disease (SD) (defined according to iRANO criteria)
BORR in CR | From date of enrollment to week 58
  Considering the best observed response for any subject, Best Overall Response Rate (BORR) is defined as the rate of complete response (CR) (defined according to iRANO criteria)
BORR in PR | From date of enrollment to week 58
  Considering the best observed response for any subject, Best Overall Response Rate (BORR) is defined as the rate of partial response (PR) (defined according to iRANO criteria)
BORR in SD | From date of enrollment to week 58
  BConsidering the best observed response for any subject, Best Overall Response Rate (BORR) is defined as the rate of stable disease (SD) (defined according to iRANO criteria)
Safety (AE) | Throughout study completion for each patient, a maximum of 58 weeks for each patient
  Safety of administration of L19TNF, through an assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Safety (SAE) | Throughout study completion for each patient, a maximum of 58 weeks for each patient
  Safety of administration of L19TNF, assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Safety (DILI) | Throughout study completion for each patient, a maximum of 58 weeks for each patient
  Evaluation of possible Drug Induce Liver Injury, caused by L19TNF, assessed by Common Toxicity Criteria (version 5.0, CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Weiss, PhD, MD, Principal Investigator — Universitatspital Zurich - Klinik fur Neurologie & Hirntumorzentrum
Locations (1):
- UniversitatSpital USZ, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No